CLINICAL TRIAL: NCT00694512
Title: Ghrelin Regulation and Structure: Effect of Diet Composition on Ghrelin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Jonathan Q. Purnell, OHSU - Center for the Study of Weight Regulation
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: eIRB 3224; OCTRI 1048 (Other: Oregon Clinical and Translational Research Institute); eIRB #3224 (Other: OHSU Institutional Review Board)
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Fat-Restricted; Diet, High-Fat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): low fat diet for two weeks.
  Interventions: Dietary Supplement: Low fat diet
- 2 (Active Comparator): High fat diet for two weeks followed by blood sampling.
  Interventions: Dietary Supplement: High fat diet
- 3 (Active Comparator): Medium Chain Triglyceride diet
  Interventions: Dietary Supplement: MCT diet

INTERVENTIONS:
Dietary Supplement: Low fat diet — 20% fat diet
  Arms: 1
Dietary Supplement: High fat diet — 40% fat diet
  Arms: 2
Dietary Supplement: MCT diet — Medium chain triglyceride diet
  Other Names: Medium chain triglyceride diet
  Arms: 3

SUMMARY:
The purpose of this study is to learn more about how diet affects the hormone ghrelin. Ghrelin is made in the stomach and causes appetite to increase. Learning about ghrelin will help the investigators understand more about obesity.

DETAILED DESCRIPTION:
Control subjects will be provided 3 different diets for 2 weeks each. At the end of each diet period participants will be admitted to OHSU Clinical Translation Research Center (CTRC) for blood sampling every 30 minutes for 13.5 hours, to measure levels of hormones. Participants will also have a DXA scan to measure body composition.

PWS subjects will have one admission after eating a standardized diet prepared by caregivers for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Weight stable for at least 3 months.
* At lifetime maximal body weight.

Exclusion Criteria:

* Actively losing weight by diet or exercise.
* Smokers.
* Alcohol consumption > 2 drinks per day.
* Exercise > 30 minutes 3 times a week.
* Prescription drug use (except birth control pills, vitamins, or minerals).
* Type 2 diabetes.
* Heart disease, cancer, malabsorptive states, or chronic infections that would affect body weight.
* Weight > 300 lbs (exceeds the weight limit of the DEXA machine).
* Hemoglobin < 12.0 g/dL for women, < 13.5 g/dL for men

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary outcomes for aim 1 are the suppression of total and acylated ghrelin from peak fasting (highest value) level to nadir (lowest level) during the 4 hours after each meal, comparing the obese to the lean subjects. | every 8 weeks

SECONDARY OUTCOMES:
Area-under-the-curve measurements during the 12 ½ hours of testing for ghrelin and other nutrient and gut-peptides, including glucose, insulin, PYY3-36, and active GLP-1. | Every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Q. Purnell, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States